CLINICAL TRIAL: NCT04196946
Title: Comparison of Bupivacaine-Fentanyl and Bupivacaine-Alfentanil Used Intrathecally in Laparoscopic Appendectomy Surgery
Brief Title: Use of Intrathecal Analgesia in Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Mehtap Balcı, Anesthesiology and Reanimation Specialist, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013/512
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia; Analgesia
Keywords: intrathecally fentanyl; alfentanil; visual pain scale; analgesia
MeSH Terms: conditions — Agnosia | interventions — Fentanyl; Alfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): 25 mcg fentanyl intrathecally
  Interventions: Drug: 25 mcg fentanyl
- Group II (Experimental): 250 mcg alfentanil intrathecally
  Interventions: Drug: 250 mcg alfentanil

INTERVENTIONS:
Drug: 25 mcg fentanyl — Before operation each patient was informed about the use of patient controlled analgesia system and visual pain scale (VPS) for pain scoring. In operating room all patient was monitored using electrocardiography (ECG), noninvasive blood pressure. Before spinal anesthesia 10-15 ml/kg intravenous serum saline infusion was started. Group I received 10 mg hyperbaric bupivacaine (2 cc) and 25 mcg fentanyl (0.5 cc).
  Other Names: fentanyl
  Arms: Group I
Drug: 250 mcg alfentanil — Before operation each patient was informed about the use of patient controlled analgesia system and visual pain scale (VPS) for pain scoring. In operating room all patient was monitored using electrocardiography (ECG), noninvasive blood pressure. Before spinal anesthesia 10-15 ml/kg intravenous serum saline infusion was started. Group II received 10 mg hyperbaric bupivacaine (2 cc) and 250 mcg alfentanil (0.5 cc) intrathecally.
  Other Names: alfentanil
  Arms: Group II

SUMMARY:
Acute appendicitis which is the most common cause of acute abdominal pain, is an acute inflammation of appendix vermiformis. Appendectomy operations can be performed as laparoscopic and open surgery. Addition of opioids to intrathecal local anesthetics to improve the quality of preoperative analgesia is an increasingly used method in recent years. The aim of this study is to compare bupivacaine-fentanyl and bupivacaine-alfentanil which are used intrathecally to create motor and sensory block. 50 volunteer patients who were diagnosed as appendicitis by laboratory tests and clinical diagnostic methods in general surgery clinic and classified as American Society of Anesthesiologists Classification I-II (ASA Class I-II) aged between 20-60 years scheduled for laparoscopic appendectomy operation, were included in this study. The patients were randomly assigned into two groups, Group I and Group II. Patients received spinal anesthesia with either 10 mg heavy bupivacaine (2 cc)+25 mcg fentanyl (0.5 cc) intrathecally (Group I, n=25) or 10 mg heavy bupivacaine (2 cc)+250 mcg alfentanil (0.5 cc) intrathecally (Group II, n=25).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who will undergo laparoscopic appendectomy operation and volunteer to participate in the study were included.

Exclusion Criteria:

* Individuals who meet the criteria but are not volunteers
* Previously underwent appendectomy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2015-09-02 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Patients diagnosis with appendicitis | With the completion of laparoscopic appendectomy operation, average 30 minutes to 1 hour
  50 volunteer patients diagnosis with appendicitis by laboratory tests and clinical diagnosis methods in general surgery clinic, aged 20-60 years with American Society of Anesthesiologists Classification I-II (ASA I-II) without contraindication for spinal anesthesia, scheduled for laparoscopic appendectomy operation were included. The patients were randomly assigned into two group.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Balcı, M.D., Principal Investigator — Nigde Omer Halisdemir University

IPD SHARING:
Plan to Share IPD: No